CLINICAL TRIAL: NCT01494025
Title: Identification of Muscle-specific Biomarkers of Fatty Acid Beta-oxidation
Acronym: FL-68
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, Davis (Other); University of Alabama at Birmingham (Other); University of Ottawa (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200816512; R01DK078328 (NIH)
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Obesity
Keywords: Diabetes; Pre-diabetes; Obese
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Glucose Intolerance | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diet and Exercise (Experimental)
  Interventions: Behavioral: Diet and Exercise

INTERVENTIONS:
Behavioral: Diet and Exercise — Subjects underwent a diet regimen targeted to elicit a 10% weight loss. Diets were designed based on the US Dietary Guidelines with caloric deficits individualized for each subject. Aerobic exercise was monitored over approximately 14 weeks, several times per week, to elicit significantly increased VO2max.

SUMMARY:
Elevated fat levels within skeletal muscle cells (intramyocellular lipids) are highly correlated with muscle and whole-body insulin resistance, and more prevalent in obesity. The molecular links and metabolic shifts driving this association remain open to debate, but notably, reduced muscle mitochondrial fatty acid (FA) ß-oxidation is more prevalent among insulin-resistant/diabetic persons. Therefore, discovery of biomarkers reflective of the status of an individual's muscle FA ß-oxidation activity or capacity would have tremendous prognostic and diagnostic value in terms of diabetes. Furthermore, characterization of metabolites associated with muscle mitochondrial fat metabolism should uncover candidate signaling factors which tie FA ß-oxidation to insulin signaling. The investigators propose to identify, for the first time, specific biomarkers of muscle FA ß-oxidation using multiple metabolomic analytical platforms to compare metabolite profiles in samples derived from biological systems displaying disparate muscle fat combustion. The current experiment will test whether plasma metabolites and/or metabolite signatures that track efficient muscular FA ß-oxidation can be experimentally increased in obese, insulin-resistant subjects via a diet-exercise regimen designed to improve muscle fitness and FA combustion.

DETAILED DESCRIPTION:
The investigators will use several comprehensive state-of-the-art metabolite analysis platforms to test the hypothesis that specific systemic metabolites or metabolite signatures correlate with myocellular fatty acid combustion. The investigators will then determine whether said metabolites do in fact reflect metabolic health status as predicted, by determining whether profiles are altered in obese subjects whose insulin sensitivity and muscle FA ß-oxidation is improved through aerobic exercise and dietary intervention. Specifically, this study is investigating the usefulness of metabolomic profiles reflective of muscle fat combustion in predicting metabolic health changes following diet & exercise intervention in obese subjects. The investigators hypothesize that biomarkers reflective of normal, efficient muscle ß-oxidation will be increased, and markers indicative of poor muscle fat combustion reduced, in a cohort of sedentary obese subjects after undergoing a 4 month diet-exercise protocol that will increase muscle fitness and improve insulin action.

In anticipation of 16 subjects completing the study, up to 20 obese female subjects will be recruited from the Davis and Sacramento areas and asked to participate in a weight loss regimen involving caloric restriction (reduction of ~25% of typical caloric intake, with rotating 7-day menus based on nutrient compositions reflective of the U.S. Dietary Guidelines) and regular aerobic exercise designed to target a 10% weight loss over 4 months (Goodpaster et al.,Diabetes 52: 2191-97, 2003). Volunteers to be included in this study will have the following characteristics: age 30-50, BMI between 30-34.9 with stable self-reported body weight over the last 6 mos., sedentary (not participating in a regular exercise program, typical planned exercise ≤30 min. per week assessed by pre-screening telephone questionnaire), non-smoker, no clinical signs of infection (i.e., no fever, CBC wnl), no personal history of cardiovascular disease, no clinically-significant elevations in blood pressure, or diabetes, no regular medications (except oral contraceptives, allergy meds) or drug abuse. These initial studies will involve women only in order to (a) reduce potential sex-related metabolite variability and (b) to better match subject characteristics in previous studies. Each subject will serve as her own control, with changes in metabolite profiles following intervention calculated for each individual. Post-absorptive insulin and glucose measurements will be made to estimate insulin sensitivity by HOMA, and patterns following an OGTT pre- and post-treatment used to assess the insulin sensitivity index using the method of Matsuda et al. (Matsuda & DeFronzo, Diabetes Care 22:1462-70, 1999). Individual changes in HOMA and insulin sensitivity values comparing pre- and post-intervention periods will be considered to be indicative of changes in insulin action. An acute exercise protocol to elicit muscle work will be carried out over 20 min. to increase metabolic flux of FA in muscle, a strategy designed to enrich the plasma with muscle metabolites. Differences in outcome variables will be tested by repeated-measures ANOVA to determine significance of fitness intervention exercise bout, and intervention exercise bout interactions.

Screening: After signing the Consent Form, an initial fasting blood draw (up to 20 mL) and vital signs will be taken to ensure potential subjects meet the clinical criteria. Height and weight will be determined and interviews conducted to evaluate whether they meet the aforementioned criteria. Body weight will be measured to the nearest 0.1kg with subjects wearing light-weight surgical scrubs. Height will be measured to the nearest 0.1cm using a wall-mounted, Ayrton Stadiometer Model S100 (Ayrton Corporation, Prior Lake, MN). Body Mass Index (BMI) will be calculated as kg/m2. Waist circumference will be measured in the standing position, with measurements obtained midway between the lateral lower rib margin and the iliac crest. The measurement will be taken mid-exhalation, and the average of two readings will be recorded. Hip circumference will be measured at the maximum protuberance of the buttocks. An additional 5 mL of blood will be drawn 2 hours after subjects consume a drink containing a 75 g dose of sugar (an abbreviated oral glucose tolerance test) in order to evaluate insulin sensitivity. A Baecke questionnaire will be used to assess physical activity level to be used in DRI calculations of maintenance calories for the pre-intervention lead-in. To minimize variability in our outcome measures that may be introduced by menstrual cycle hormonal shifts, we will endeavor to maintain consistency by evaluating subjects during the follicular phase of the menstrual cycle (as estimated by cycle records for each woman), preferably beginning on day 4 of the menstrual cycle. Subjects on birth control medication will also preferably be evaluated on day 4 of their menstrual cycle. Subjects will be given a calendar and instructions to record their menstrual cycles throughout the study. Eligible subjects will be asked to visit the WHNRC several times, as follows:

Test Week 1: On day 4 of their menstrual cycle, subjects will come to the clinic for the beginning of Test Week 1. Each day subjects will be given prepared meals to be eaten at the WHNRC, or packed to go along with final preparation instructions. During the test week subjects will receive meals and snacks for a 7 day menu prepared by the WHNRC Metabolic Kitchen and based on U.S. Dietary Guidelines and prescribed to maintain stable body weight. Volunteers will be provided with a daily multivitamin supplement study and will be required to refrain from taking personal dietary supplements or vitamins during the study. This is designed to ensure a similar nutritional profile across all subjects, prior to obtaining biofluids for metabolomic analysis to minimize physiological variability. Subjects will be weighed daily during Test weeks 1 and 2 to ensure body weight maintenance and diet prescriptions adjusted if necessary. During this test week each subject will participate in an instruction session regarding the diet and diet compliance provided under the guidance of a registered dietitian. This instruction may be done individually or in a group setting. Each individual's diet (based on the U.S. Dietary Guidelines) and exercise plan will be designed to elicit a target of 10% body weight loss and to improve fitness over the 16 week intervention period. Test Week 2: Test week 2 duplicates Test Week 1. Subjects will be scheduled based on predictions from their menstrual calendars. This might mean that subjects will continue exercising for additional days in order to coincide with menstrual day 4 when diet is provided and testing begins. The acute exercise will be a 40-50% of the Test week 1 VO2max.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 30-50
* menstruating with regularity
* BMI between 30- 37.5 with stable body weight (<5% change) over last 6 mos
* waist to hip ratio >0.9
* sedentary lifestyle (typical exercise < 30 min. per week)
* non-smoker
* evidence for pre-diabetes (hyperinsulinemia and/or blood glucose > 100 < 126 mg/dl)

Exclusion Criteria:

* any clinically significant abnormal laboratory values
* any clinical signs of infection (i.e., fever)
* any chronic diseases
* any personal history of cardiovascular disease
* clinically-significant elevation in blood pressure (≥130/85)
* diabetes or other chronic disease
* any regular medications or drug abuse
* pregnancy or lactation

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in VO2max | Week 1 vs. Week 16
  Overnight fasted subjects will start the test at a low cycle ergometer resistance level and encouraged to maintain a steady rate of pedaling, and resistance will increase at 2-min intervals until volitional fatigue. Indirect calorimetry will be used to measure VO2 and CO2 continuously during the exercise test. Subjects will receive a pre-test ECG, breath volume test and medical exam to assure the subject has no underlying medical problems that would put them at an undue risk during the exercise tests.
Change in Body Composition (BODPOD) | Week 1 vs. Week 16
  Body fat mass and fat-free mass will be measured using the BOD POD. Subjects will be asked to change into a provided form-fitting swimsuit or single layer compression shorts and single layer jog bra for women. Subjects will also be asked to wear a provided swim cap to compress the hair on their head. After measuring height and weight, they will sit comfortably in the BOD POD and limit their movement while breathing normally. During the last section of the test subjects will be asked to breathe into a tube and give three puffs when indicated by the computer screen.
Change in Insulin Sensitivity | Week 1 vs. Week 16
  OGTT (oral glucose tolerance test) A standard oral 75 g glucose tolerance test (OGTT) will be administered and the insulin sensitivity index calculated as per Matsuda and DeFronzo. For screening a blood sample will be taken after 2 hours. For the test week, blood samples will be taken at 0, 15, 30, 60, 90, and 120 min post-glucose ingestion (up to 8 mL of blood will be obtained/timepoint).
Change in Metabolite Profiling and Metabolomics | Week 1 vs. Week 16
  EDTA plasma from overnight fasted subjects and samples derived from exercise tests obtained in the pre-intervention and post-intervention test weeks will be analyzed. Samples will be analyzed using several mass spec based metabolomics platforms. Exercise samples are derived from subjects undergoing 30-minutes of submax exercise (45% VO2max) collected every 5 minutes, plus samples collected during a 20-minute cool-down phase.
Change in Body Composition (DXA) | Week 1 vs. Week 16
  Body fat mass and fat-free mass will be measured by DXA using a whole body scan. The scan will be performed at the beginning of the study and after the diet and exercise intervention. Our technical staff at WHNRC is trained and certified in the DXA method. The volunteer will wear light-weight surgical scrubs. The scan time takes no longer than 30 minutes to complete, with a radiation exposure less than 0.1 mrem. As subjects will be menstruating during the test week, there is no risk to a developing fetus. A pregnancy test will be offered but not required.
Change in Body Weight | Week 1 vs. Week 16
  Body weights are measured on a calibrated scale approximately on a weekly basis throughout the study, and daily during pre-intervention Test Week 1 and post-intervention Test Week 2.

CONTACTS AND LOCATIONS:
Overall Officials: Sean H Adams, PHD, Principal Investigator — University of California, Davis
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- See also: Western Human Nutrition Research Center, Davis, CA — https://www.ars.usda.gov/pacific-west-area/davis-ca/whnrc/